CLINICAL TRIAL: NCT02721004
Title: Documentation of the Efficacy and Safety of RoActemra in the Treatment of Rheumatoid Arthritis
Brief Title: Efficacy and Safety Study of RoActemra (Tocilizumab) in Participants With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22551
Record Dates: First submitted 2016-03-02; First posted 2016-03-28 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-07

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; RoActemra; Tocilizumab
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Rheumatoid arthritis participants: Rheumatoid arthritis participants receiving tocilizumab intravenous infusion every 4 weeks according to product label/per standard practice for a maximum of 12 months will be observed in this study.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab administered as an intravenous infusion every 4 weeks according to product label/per standard practice for a maximum of 12 months will be observed in this study.
  Other Names: RoActemra

SUMMARY:
This is an open-label, non-interventional study to evaluate efficacy and safety in rheumatoid arthritis participants receiving tocilizumab as per the product label.

ELIGIBILITY:
Inclusion Criteria:

- Participants with rheumatoid arthritis receiving tocilizumab as per product label

Exclusion Criteria:

- No specific exclusion criteria were specified for this non-interventional trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with rheumatoid arthritis will be enrolled in this trial.
Sampling Method: Non-Probability Sample
Enrollment: 592 (Actual)
Dates: Start 2009-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Disease Activity Score Based on 28-joints Count (DAS28) | Month 12
Simplified Disease Activity Index (SDAI) Score | Month 12
Clinical Disease Activity Index (CDAI) Score | Month 12
Percentage of Participants Achieving American College of Rheumatology (ACR) Response | Month 12
Tender Joint Count (TJC) | Month 12
Swollen Joint Count (SJC) | Month 12

SECONDARY OUTCOMES:
Percentage of Participants with any Adverse Event (AE) | Up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Bludenz, Austria